CLINICAL TRIAL: NCT06698939
Title: Phase 1, First-in-human, Double-Blind, Placebo-Controlled, Single Dose Escalation Study to Evaluate the Safety, Tolerability, and Pharmacokinetics, of ORKA-001 in Healthy Participants
Brief Title: ORKA-001 in Healthy Volunteers
Acronym: ORKA-001-111
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Oruka Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: ORKA-001-111
Record Dates: First submitted 2024-11-13; First posted 2024-11-21 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Healthy Volunteers
Keywords: ORKA-001; Phase 1

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ORKA-001 (Experimental): Participants will receive subcutaneous injection of ORKA-001 at either 300 mg, 600 mg or 1200 mg.
  Interventions: Drug: ORKA-001
- Placebo (Placebo Comparator): Participants will receive a subcutaneous injection of placebo comparator.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: ORKA-001 — ORKA-001 is supplied as sterile solution to be administered by SC injection
  Arms: ORKA-001
Other: Placebo — Placebo solution to be administered at a matching volume by SC injection
  Arms: Placebo

SUMMARY:
This is a Phase 1, First-in-human Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of ORKA-001 in Healthy Participants.

DETAILED DESCRIPTION:
This is a single center, phase 1, double-blind, placebo-controlled, randomized, first-in-human (FIH), single ascending dose study evaluating the safety, tolerability, and pharmacokinetics (PK) of ORKA-001 in healthy volunteers. The study will enroll approximately 24 healthy volunteers. The ORKA-001 dose will be administered by a subcutaneous injection.

ELIGIBILITY:
Key Inclusion Criteria:

1. Healthy male or female participants
2. 18 to 65 years (inclusive) with a body mass index (BMI) 18 to 32 kg/m2
3. Willing and able to remain at the study site unit for the duration of the confinement period and return for the outpatient visit/s defined in the protocol
4. Using a highly effective method of contraception from admission through the end of the study.
5. Willing to abstain from regular, continuous alcohol use or tobacco use as per protocol

Key Exclusion Criteria:

1. Any clinically significant medical condition or finding that, in the Investigator's opinion, is likely to unfavorably alter the risk of study participation, confound study results, or interfere with the study conduct or compliance.
2. Known history of illicit drug use or drug abuse or harmful alcohol use
3. Known history of frequent tobacco or vaping use within 2 years prior to Screening
4. History of severe allergic reactions or hypersensitivity
5. Actively nursing or lactating
6. Use of investigational drug therapy within 30 days prior to enrollment
7. Unable to comply with study requirements or in the opinion of the Investigator should not participate in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-12-19 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Number and frequency of Treatment-Emergent Adverse Events [Safety and Tolerability] | Day 1 through one year
  Incidence of treatment-emergent adverse events (TEAEs) and clinically significant changes from baseline in vital signs, electrocardiograms (ECGs), clinical laboratory parameters, and physical examinations.

SECONDARY OUTCOMES:
Maximum observed serum concentration of ORKA-001 | Day 1 through one year
  CMax of ORKA-001
Time to CMax (TMax) of ORKA-001 | Day 1 through one year
  TMax of ORKA-001
Area Under the Serum Concentration-Time Curve (AUC) of ORKA-001 | Day 1 through one year
  Area under the curve from the time of dosing to infinity (AUC0-inf)
Terminal elimination half-life (T1/2) | Day 1 through one year
  T1/2 of ORKA-001

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Breitschwerdt, Study Director — Oruka Therapeutics, Inc.; Principal Investigator, Principal Investigator — Oruka Therapeutics Investigative Site
Locations (1):
- Oruka Therapeutics Investigative Site, Christchurch, New Zealand